CLINICAL TRIAL: NCT06165692
Title: The Use of Platelet-rich-fibrin in Lower Third Molar Surgery: a Split-mouth Randomized Clinical Trial
Brief Title: The Use of Platelet-rich-fibrin in Lower Third Molar Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amerigo Giudice (Other)
Responsible Party: Sponsor-Investigator, Amerigo Giudice, Professor, University Magna Graecia
Organization: University Magna Graecia (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2/2023
Record Dates: First submitted 2023-11-15; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Facial Swelling; Tooth Position Anomalies; Tooth, Impacted; Tooth Extraction Status Nos; Tooth Avulsion
Keywords: third molar surgery; facial swelling; 3D facial swelling evaluation; PRF; tooth impacted; platelet rich fibrin
MeSH Terms: conditions — Tooth, Impacted; Tooth Avulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Placement of PRF in the post-extraction socket after third molar surgery
  Interventions: Biological: PRF
- Control Group (No Intervention): No positioning PRF in the post-extraction socket after third molar surgery

INTERVENTIONS:
Biological: PRF — Post-operative PRF placement in the post-extraction socket after third molar surgery
  Arms: Test Group

SUMMARY:
The present study aims to analyze the effect of PRF (Platelet-rich-fibrin) in terms of facial swelling, trismus and pain after surgical removal of mandibular third molar (M3M) in a split-mouth randomized controlled clinical trial.

DETAILED DESCRIPTION:
The present study aims to analyze the effect of PRF (Platelet-rich-fibrin) in terms of facial swelling, trismus and pain after surgical removal of mandibular third molar (M3M) in a split-mouth randomized controlled clinical trial. Facial swelling will be assessed using an innovative three-dimensional digital technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 32 years who required both M3M extractions were recruited
* Good health status
* Indication to surgical extraction of both M3M
* Complete root formation
* Surgical risk level classified as "Conventional" or "Moderate" according to Daugela et al. classification

Exclusion Criteria:

* Person under the age of 18 or over 32
* Allergy or contraindications to administration of corticosteroids
* Acute infection in any of the teeth to be extracted
* Patients with chronic liver disease, diabetes, immune system dysfunction, or haematological disease
* Pregnancy or breastfeeding
* History of treatment with antiresorptive drugs
* Chronic kidney disease

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Facial swelling qualitative analysis | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of PRF in reducing facial swelling using qualitative three-dimensional analysis (measured by colorimetric variation given by the overlapping volumes) .
Facial swelling quantitative analysis - volumetric differences | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of PRF in reducing facial swelling using quantitative three-dimensional analysis ( volumes measured in cm3) .
Facial swelling quantitative analysis - linear differences | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of PRF in reducing facial swelling using quantitative three-dimensional analysis (linear differences measured in cm2) .

SECONDARY OUTCOMES:
Trismus analysis | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To assess the effects of PRF administration on trismus (measured in cm)
Pain analysis with Visual analogue scale (VAS) | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To assess the effects of PRF administration on pain (measured by VAS-score from 0 to 10 point, with 10 as the worst outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Magna Graecia University of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No